CLINICAL TRIAL: NCT05201157
Title: The Effect of Acupressure on Postpartum Fatigue in Women Who Had Cesarean Delivery: A Randomized Controlled Study
Brief Title: Nonpharmacological Method and Postpartum Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: resmiye kaya odabaş (Other)
Responsible Party: Sponsor-Investigator, resmiye kaya odabaş, Principal Investigator, Aydin Adnan Menderes University
Organization: Aydin Adnan Menderes University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Resmiye-02
Record Dates: First submitted 2022-01-07; First posted 2022-01-21 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Fatigue
Keywords: postpartum fatigue; postpartum; fatigue; acupressure
MeSH Terms: conditions — Fatigue | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupressure group (Active Comparator): Acupressure will be applied to ST36, LI4 and SP6 points.The Introductory Information Form will be filled in by the researcher and the Visual Similarity Scale for Fatigue will be filled by women once on the post-op 0th day and once on the post-op 2nd day, a total of 2 times.
  Interventions: Other: acupressure group
- Control Group (Active Comparator): No application will be made to this group, and the Introductory Information Form will be filled in by the researcher and the Visual Similarity Scale for Fatigue will be filled in 2 times in total, once on the post-op 0th day and once on the post-op 2nd day.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: acupressure group — A suitable environment will be prepared for mothers in terms of warmth and light, where privacy can be protected. The application points will be determined with the acu-point device by choosing the most comfortable position of the mother, leaving the application points exposed. The most preferred points ST36, LI4 and SP6 were selected from the points reported to affect lactation by reviewing the literature on the points to be compressed. Acupressure will be applied to points (bidirectional, right and left) for 2 minutes for a total of 6 minutes. Light pressure will be applied with the thumb of the practitioner's hand. Immediately after applying pressure for 2 minutes for each point, it will be moved to the other point in the symmetrical region and the application will be made without interruption. While practicing, the researcher will control the time using a digital wrist watch with a stopwatch
  Arms: Acupressure group
Other: Control Group — No application will be made. The mothers in this group will fill in the Visual Similarity Scale for Fatigue twice, once between 8-12 hours post-op and once on the post-op 2nd day.
  Arms: Control Group

SUMMARY:
Postpartum fatigue is common in women after cesarean section and it affects the woman and the baby. Many noninvasive applications help to overcome this problem. This study was planned as a randomized controlled trial to examine the effect of acupressure on postpartum fatigue in women who had a cesarean section. The research will be carried out between August 2021 and August 2022 with mothers who have had a cesarean section at Kocaeli University Research and Application Hospital. The research will be carried out with two groups as acupressure and control group. The sample number was calculated using the G*Power 3.1.9.2 program and the acupressure group: 60 and the control group: 60. In order to increase the analysis power, the number of people for each group was taken as 65 (n=130). It is planned to collect the data with the Descriptive Information Form and the Visual Similarity Scale for Fatigue. Acupressure will be applied to the mothers in the acupressure group once, once on the post-op day 0, twice on the post-op 1. day and once on the post-op 2. day, for a total of 4 times for six minutes, and no application will be made to the control group. Fatigue will be assessed with the Visual Similarity Scale for Fatigue before administration on post-op day 0 and after administration on post-op day 2. The data of the research will be evaluated using the Statistical Package for the Social Sciences 22.0 program. In the evaluation of the data; descriptive statistics will be given as percentage, arithmetic mean±standard deviation, median and minimum-maximum values. Independent two-sample t-test will be used for normally distributed variables, and Mann-Whitney U test for non-normally distributed variables. Pearson Correlation test will be applied to determine the relationship between the fatigue severity of the experimental group and the tests and to determine the relationship between the tests. Statistical significance level will be accepted as p<0.05.

DETAILED DESCRIPTION:
Aim: The aim of this study is to determine the effect of acupressure on postpartum fatigue in women who had cesarean section.

Hypotheses:

H0: There is no difference in fatigue between the acupressure group and the control group in women who had cesarean section.

H1: There is a difference in fatigue between the acupressure group and the control group in women who had a cesarean section.

This study was designed as a randomized controlled experimental study. The study was carried out in "Kocaeli University Research and Application Hospital" and "Health Sciences University Derince Training and Research Hospital" obstetrics service between August 2021 and August 2022 planned to be carried out.

The population of the research will be the mothers who gave birth by cesarean section in "Kocaeli Provincial Health Directorate Health Sciences University" and "Health Sciences University Derince Training and Research Hospital- Alikahya Campus". To determine the sample size in the study, it was calculated based on the study conducted to examine the effect of meridian acupressure massage on body composition, edema, stress and fatigue in postpartum women. The sample size of the study was calculated using the G*Power 3.1.9.2 program, and the mean, standard deviation and sample number values of the fatigue score after the intervention in the related article were taken into account in calculating the effect size. The mean and standard deviation values of the fatigue score after the intervention in the experimental group were 49.95±11.43 and n=19. In the control group, the mean and standard deviation values of the fatigue score were 58.55±20.25 and n=20. The effect size was calculated as 0.52 by using the mean, standard deviation and sample number values of the related article. 95% confidence (1-α), 80% test power (1-β), d=0.52 effect size, the minimum number of samples to be taken in each group according to the independent samples t-test result is 60, a total of 120 cases to be examined. required. In order to increase the analysis power, n=65 will be taken for each group in the study (experimental group: 65 and control group: 65). Pregnant women in the acupressure group and control group will be stratified in terms of age and homogeneous distribution of the groups will be ensured. In which group the women included in the study will take place will be determined from the website of the random number generation program "Random Team Generator", and they will be divided into two groups. Thus, each woman's number and group number will be determined and recorded.

Introductory Information Form: This form was created by researchers based on the literature. The form consists of a total of 18 questions questioning the socio-domographic and obstetric characteristics of women and their general health status.

Visual Similarity Scale for Fatigue: The scale consists of 18 items, including fatigue (items 1, 2, 3, 4, 5, 11, 12, 13, 14, 15, 16, 17, 18) and energy (items 6, 7, 8, 9, 10). ) consists of two sub-dimensions. The scale consists of 10 cm horizontal lines with positive statements on one end and negative statements on the other. While the items of the fatigue sub-dimension move from positive to negative, the items of the energy sub-dimension are in the opposite order. The lowest score obtained in the fatigue sub-dimension is 0, and the highest score is 130. In the energy sub-dimension, scores are calculated in the range of 0-50 points. The high score of the fatigue sub-dimension and the low score of the energy sub-dimension indicate that the severity of fatigue increases. In the validity and reliability study of the scale, it was reported that the Cronbach's α internal consistency coefficient was 0.9 for the 13-item fatigue subscale, 0.74 for the 5-item energy subscale, and the correlations between all the items of the scale were significantly high. This scale will be used twice for each woman. The scale will be applied twice in both groups.Permission was obtained from the author for the use of the scale.

Pre-Application In order to assess whether the questions have been understood, a preliminary study will be conducted with five mothers before starting the study. As a result of the evaluation, it will be evaluated whether there is a need for editing in the data forms and adjustments will be made. Those included in the preliminary study will not be included in the sample group.

Data Collection After obtaining the permissions of the ethics committee and the institution, the study can be performed by going to the institutions and performing a cesarean section between the first 8-12 hours on the 0th postoperative day. Mothers who are between working hours will be welcomed. Mothers who meet the research criteria will be informed about the purpose, content and method of the research and those who want to participate in the research will be determined.

After cesarean section for women;

* Post-operative between 8-12. hours (1 time),
* Post-operative 1st day (2 times),
* Acupressure will be applied once on the 2nd post-op day 4 times in total, .

Visual Similarity Scale for Fatigue by women;

* Post-operative between 8-12. hours 1 time (before application),
* Once on the 2nd post-op day. It will be filled 2 times in total.

Acupressure Application Technique: A suitable environment will be prepared for mothers in terms of warmth and light, where privacy can be protected. The application points will be determined with the acu-point device by choosing the most comfortable position for the mother, leaving the application points exposed. The most preferred points Stomach (ST) 36, Spleen (SP) 6 and Large Intestine (LI4) were selected from the points reported to affect lactation by examining the literature on the points to be applied. Acupressure will be applied to at all point (bidirectional, right and left) for 2 minutes for a total of 6 minutes. Light pressure will be applied with the thumb of the practitioner's hand. Immediately after applying pressure for 2 minutes for each point, it will be moved to the other point in the symmetrical region and the application will be made without interruption. While practicing, the researcher will control the time using a digital wrist watch with a stopwatch.

The assistant researcher received acupressure training on 13.05.2021 and the principal researcher also has acupressure training.

Acupressure Application Points:

ST 36 point: It can also be used for gastrointestinal symptoms such as respiratory distress, fatigue, nausea-vomiting, slowing of bowel movements, bloating, loss of appetite, dizziness and insomnia. By stimulating the spleen and stomach. the amount of energy going to the lungs is increased.

SP6 poin: This point, which is generally used for urological and pelvic problems, menstrual pain and insomnia, is also preferred in various studies to reduce fatigue.

LI4: Although this area is generally used for face, head and toothache, it is also a frequently preferred area to increase alertness and reduce fatigue.

The data of the study will be evaluated using the Statistical Package for the Social Sciences (SPSS) 22.0 program. All data will first be evaluated with the Kolmogorov-Smirnov test for conformity to normal distribution, and then analyzed according to conformity to normal distribution. For descriptive statistics, percentages will be used in general, arithmetic mean±standard deviation for those suitable for normal distribution, median and minimum-maximum values for those that do not fit. Comparisons between groups for numerical variables of socio-demographic and clinical characteristics will be made with an independent two-sample t-test for normally distributed variables, and Mann-Whitney U test for non-normally distributed variables. Pearson Correlation test will be applied to determine the relationship between the fatigue severity of the experimental group and the tests and to determine the relationship between the tests. Statistical significance level will be accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18-35,
* Birth after 36th gestational week,
* Multiparous
* Caesarean section with regional anesthesia,
* Mobilized,
* Not having any health problems (Hypertension, tuberculosis, HIV, cancer, psychological disorders, etc.),
* Does not have any problems preventing communication,
* At least primary school graduate,
* Able to speak and understand Turkish,
* Volunteer women who agreed to participate in the study

Exclusion Criteria:

* Having postpartum complications (bleeding, embolism, eclampsia, infection, etc.),
* Having a hemoglobin level of less than 9 g/dl and a hematocrit level of less than 30%,
* Having a body mass index of 40 and above,
* Covid-19 test positive,
* Having twin babies,
* The baby is in the neonatal intensive care unit,
* Having been diagnosed psychologically (such as depression) before,
* Women who do not want to participate in the research will be excluded from the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2021-08-12 (Actual); Primary Completion 2022-01-09 (Actual); Study Completion 2022-03-13 (Actual)

PRIMARY OUTCOMES:
Visual Similarity Scale for Fatigue | This scale will be filled by mothers between 8-12 hours after cesarean section.
  The scale consists of 18 items, including fatigue (items 1, 2, 3, 4, 5, 11, 12, 13, 14, 15, 16, 17, 18) and energy (items 6, 7, 8, 9, 10). ) consists of two sub-dimensions. The scale consists of 10 cm horizontal lines with positive statements on one end and negative statements on the other. The lowest score obtained in the fatigue sub-dimension is 0, and the highest score is 130. In the energy sub-dimension, scores are calculated in the range of 0-50 points. The high score of the fatigue sub-dimension and the low score of the energy sub-dimension indicate that the severity of fatigue increases.
Visual Similarity Scale for Fatigue | This scale will be filled in by the mothers between in postoperative period on 2.days at 08.00-16:00 am]
  The scale consists of 18 items, including fatigue (items 1, 2, 3, 4, 5, 11, 12, 13, 14, 15, 16, 17, 18) and energy (items 6, 7, 8, 9, 10). ) consists of two sub-dimensions. The scale consists of 10 cm horizontal lines with positive statements on one end and negative statements on the other. The lowest score obtained in the fatigue sub-dimension is 0, and the highest score is 130. In the energy sub-dimension, scores are calculated in the range of 0-50 points. The high score of the fatigue sub-dimension and the low score of the energy sub-dimension indicate that the severity of fatigue increases.

CONTACTS AND LOCATIONS:
Overall Officials: Resmiye Kaya Odabaş, Ress. Ass., Principal Investigator — Kocaeli University; Yasemin Sökmen, Instructor, Study Chair — Ondokuz Mayıs University; Ayten Taşpınar, Prof Doctor, Study Chair — Aydin Adnan Menderes University
Locations (1):
- Aydın Adnan Menderes University, Efeler, Aydın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No